CLINICAL TRIAL: NCT04179123
Title: 3D Printing of Positive Airway Pressure (PAP) Therapy Masks: a Single Site Pilot and Feasibility Study
Acronym: 3DPiPPIn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 18/0052
Record Dates: First submitted 2019-11-15; First posted 2019-11-27 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Two phase feasibility trial:
  Phase 1: 10 healthy subjects Phase 2: 10 patients already on PAP therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Experimental): Conventional and customised PAP interfaces
  Interventions: Device: Customised PAP interfaces
- Patients (Experimental): Conventional and customised PAP interfaces
  Interventions: Device: Customised PAP interfaces

INTERVENTIONS:
Device: Customised PAP interfaces — Customised PAP interfaces

SUMMARY:
This study is a single site pilot and feasibility study. We propose that 3D printing could be used to create customised masks for patients requiring Positive Airway Pressure (PAP) therapy. We hypothesise that the use of this technology may result in; improved compliance with therapy, increased comfort, reduced side effects, increased quality of life and reduced healthcare costs.

DETAILED DESCRIPTION:
Stage 1:

10 health participants. subjects will be asked to attend for a mask fitting using off the shelf standard mask stock. They will then be trialed on PAP therapy (breathing machine) for 10 minutes. Mask leak, skin reactions and comfort scores will be assessed.

Subjects will then attend for 3D printing of a mask. Following the production of the 3D mask, repeat measurements with the 3d mask on PAP therapy will be taken.

If all healthy subjects complete the trial without any serious adverse events, then the second phase of the study with patients will commence.

Stage 2:

Patients with an established diagnosis of sleep disordered breathing with known mask concerns will be recruited from the Royal Free London NHS Foundation Trust (RFL) Sleep and Ventilation Service. Subjects will be asked to attend for a mask fitting using their existing mask standard stock and will be trialed on PAP therapy (breathing machine) for 10 minutes. Mask leak, skin reactions and comfort scores will be assessed. Any side effects will be documented via photographs. The number and cost of previous masks used since starting PAP therapy (breathing machine) will be also be recorded.

Patients will then attend for 3D printing of a mask and repeat measurements with the 3D mask on 10 minutes of their usual PAP therapy will be taken. If there are no serious adverse events/reactions during the PAP trial with the 3D printed mask patients will go on to have a one-night trial on PAP therapy as per their normal PAP (breathing machine) regime. If there are no adverse events or reactions during the one-night trial then patients will proceed to a further four nights of trial with the 3D printed mask. A comparison of scores will be made with standard and 3D printed masks.

ELIGIBILITY:
Healthy:

Inclusion Criteria:

* Members of staff working at Royal Free London NHS Foundation Trust

Exclusion Criteria:

* Staff with known sleep disordered breathing. Staff with suggestion of sleep disordered breathing on the STOP Bang and Epworth Sleepiness Score screening tools

Patients

Inclusion Criteria:

* Patients will be recruited from the existing sleep and ventilation database at RFL. Patients with an established diagnosis of sleep disordered breathing with known interface concerns will be recruited. Patients who have been identified as having problematic interface concerns resulting in mask leak, poor mask fit, pressure ulcers and reduced effectiveness of PAP therapy

Exclusion Criteria:

* Patients who are clinically unstable as assessed by a clinical member of the research team. Patients with evidence of active infection on clinical assessment. Patients who have dependent on their therapy for more than 16 hours in a 24 hour period. Patients with active pressure ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
To pilot the feasibility of using 3D printing technology to develop customised masks for patients receiving PAP therapy. This will be assessed through the secondary outcome measures and the Medical Research Council Complex Intervention Framework | 5 days
  Acceptability of 3D printed customised PAP masks by patients and healthcare professionals

SECONDARY OUTCOMES:
Comfort | 5 days
  Measured with self developed mask comfort questionnaire. Combination of questions answered on a Visual Analogue Scale (1-5) scale, open questions and binary questions. No overall score produced
Side effects | 5 days
  Measured with self developed mask comfort questionnaire. Combination of questions answered on a VAS scale, open questions and binary questions. No overall score produced.
  Objective assessment of skin to assess for skin reactions, graded with the EUPAP 0-4.
Mask leak | 5 days
  Measured via SD data card download. Leak a l/min as an average over 5 nights

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free London NHS foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No